CLINICAL TRIAL: NCT02491229
Title: Clinical Trial for Investigating the Effects of "Hepafast" on Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: "Hepafast" in Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: Bodymed AG (Unknown)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Stephan C. Bischoff, MD, Professor, University of Hohenheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKES HEPA V2.0
Record Dates: First submitted 2015-02-03; First posted 2015-07-07 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Obesity
Keywords: non-alcoholic fatty liver disease (NAFLD); Obesity; Hepafast
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Hepafast" (Other): This group consumes three portions of "Hepafast" and additionally 200 kcal of vegetables for two weeks. In the following ten weeks, they consume two portions of "Hepafast" and one meal which follows the instructions of the Low Glycemic and Insulinemic Diet (LOGI).
  Interventions: Other: Hepafast
- Control (Other): This group follows the instruction of the LOGI diet for the entire 12 weeks
  Interventions: Other: LOGI diet

INTERVENTIONS:
Other: Hepafast — Two weeks of Hepafast three times a day and additionally 200 kcal followed by 10 weeks of Hepafast two times a day and a meal according to LOGI diet
  Arms: "Hepafast"
Other: LOGI diet — For twelve weeks, this group eats meals according to the Low Glycemic and Insulinemic Diet (LOGI).
  Arms: Control

SUMMARY:
The purpose of this study is to investigate whether a weight reduction with "Hepafast" in combination with raw food and vegetables for two weeks followed by a meal substitution with "Hepafast" and a calorie restriction in accordance with the Low Glycemic and Insulinemic Diet (LOGI) for 10 weeks is superior regarding improvement of non-alcoholic Fatty Liver Disease (NAFLD) compared to a conventional weight reduction in accordance with the LOGI diet without use of "Hepafast" for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30-40 kg/m2
* suspected or diagnosed non-alcoholic fatty liver disease (NAFLD)

Exclusion Criteria:

* other liver diseases
* kidney failure
* pregnancy, lactation
* diabetes mellitus which is treated with insulin
* alcohol abuse
* several drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change from baseline in hepatorenal index at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.

SECONDARY OUTCOMES:
change from baseline in fatty liver index at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in the classification of non-alcoholic fatty liver disease (NAFLD) based on ultrasound at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in body weight at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in blood pressure (systolic and diastolic) at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in GGT at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in GOT at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in GPT at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in AP at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in triglycerides at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in HDL cholesterol at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in LDL cholesterol at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in fasting glucose at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in insulin at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in HbA1c at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.
change from baseline in hsCRP at two weeks, six weeks and twelve weeks after starting a defined way of nutrition | Participants will be followed for the time of twelve weeks. Examinations take place at two weeks, six weeks and twelve weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, Principal Investigator — University of Hohenheim
Locations (1):
- University of Hohenheim, Stuttgart, Germany